CLINICAL TRIAL: NCT04239677
Title: Impact of Retrograde Autologous Priming on the Coagulation Profile Assessed by Rotation Thromboelastometry (ROTEM) in Patients Undergoing Cardiac Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2019-1088
Record Dates: First submitted 2020-01-14; First posted 2020-01-27 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Cardiac Surgery; Vascular Surgery Using CPB
Keywords: retrograde autologous priming; ROTEM; Cardiac surgery; Vasculsr surgery using CPB

STUDY DESIGN:
Intervention Model Description: Prospective randomized trial with 2 parallel groups; the retrograde autologous priming group and conventional crystalloid solution-based priming group.
Who Masked: Participant, Outcomes Assessor
Masking Description: One investigator (Anesthesiologist) conducts randomized group assignment. The day of surgery, the researcher informs to surgeon, perfusionist about patient's group assignment.
  But, other researcher (ROTEM test), postoperative management do not know the patient's group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Conventional crystalloid solution-based priming
  Interventions: Procedure: Conventional crystalloid solution-based priming
- RAP (Experimental): Retrograde autologous priming
  Interventions: Procedure: Retrograde autologous priming

INTERVENTIONS:
Procedure: Conventional crystalloid solution-based priming — CPB circuit is also prepared with crystalloid solution-based priming in all participants (same as the RAP group). In this group (control group), CPB is initiated with antegrade priming (conventional priming).
  Arms: control
Procedure: Retrograde autologous priming — CPB circuit is prepared with crystalloid solution-based priming in all participants. In RAP group, retrograde autologous priming is performed by displacing the crystalloid priming volume of arterial and venous lines via passive exsanguination of native blood prior to CPB initiation.
  Arms: RAP

SUMMARY:
Cardiac surgery with cardiopulmonary bypass (CPB) is associated with an increased risk of blood transfusions. The primary setup of the CPB circuit demands a priming volume of approximately 1600 mL of crystalloid solution which leads to a relevant hemodilution. The retrograde autologous priming (RAP) procedure minimizes hemodilution by displacing the crystalloid priming volume of arterial and venous lines via passive exsanguination of native blood prior to CPB initiation, resulting in higher hematocrits and reduction of red blood cell transfusion. RAP can also minimize the dilution of coagulation factors as well as red blood cells. Thus, the investigators hypothesized that RAP could maintain better coagulatory function after CPB. In this study, the investigators investigate the impact of RAP on the coagulation profile assessed by rotation thromboelastometry (ROTEM) in participants undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 20 years of age undergoing cardiac surgery / vascular surgery using CPB

Exclusion Criteria:

* Emergency operation
* Hemoglobin concentration above 15g/dL
* Anticoagulants such as warfarin within 5 days before surgery, non-vitamin K antagonist oral
* anticoagulant within 2 days, and aspirin / clopidogrel / ticagrelor within 5 days
* Weight less than 45kg, more than 90kg
* Patients with autoimmune disease
* Patients who participated in other clinical studies that could affect prognosis
* Patients who cannot understand the informed consent (eg. Foreigner)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2020-02-06 (Actual); Primary Completion 2021-09-03 (Actual); Study Completion 2021-09-03 (Actual)

PRIMARY OUTCOMES:
Maximal Clot firmness (MCF) of Externally activated ROTEM assay (EXTEM) | 10 minutes after induction of anesthesia
  Maximal Clot firmness (MCF) of EXTEM is a ROTEM parameter representing the strength of a clot, the formation of which is triggered by an activator of extrinsic coagulation pathway.
Maximal Clot firmness (MCF) of EXTEM | 1 minutes after rewarming (during CPB)
  Maximal Clot firmness (MCF) of EXTEM is a ROTEM parameter representing the strength of a clot, the formation of which is triggered by an activator of extrinsic coagulation pathway.
Maximal Clot firmness (MCF) of EXTEM | 15 minutes after injection of protamine (after cessation of CPB for reversal of heparin)
  Maximal Clot firmness (MCF) of EXTEM is a ROTEM parameter representing the strength of a clot, the formation of which is triggered by an activator of extrinsic coagulation pathway.
  Dosage of heparin and protamine is only affected by patients' real body weight (not by ROTEM results).
  That is, in each case, the same protamine dosage applies to both groups.

SECONDARY OUTCOMES:
Clotting Time (CT) | 10 minutes after induction of anesthesia
  Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
Clotting Time (CT) | 1 minutes after rewarming (during CPB)
  Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
Clotting Time (CT) | 15 minutes after injection of protamine (after cessation of CPB for reversal of heparin)
  Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
  Dosage of heparin and protamine is only affected by patients' real body weight (not by ROTEM results).
  That is, in each case, the same protamine dosage applies to both groups.
Clot Formation Time (CFT) | 10 minutes after induction of anesthesia
  Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
Clot Formation Time (CFT) | 1 minutes after rewarming (during CPB)
  Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
Clot Formation Time (CFT) | 15 minutes after injection of protamine (after cessation of CPB for reversal of heparin)
  Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
  Dosage of heparin and protamine is only affected by patients' real body weight (not by ROTEM results).
  That is, in each case, the same protamine dosage applies to both groups.
A10 | 10 minutes after induction of anesthesia
  Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
A10 | 1 minutes after rewarming (during CPB)
  Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
A10 | 15 minutes after injection of protamine (after cessation of CPB for reversal of heparin)
  Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
  Dosage of heparin and protamine is only affected by patients' real body weight (not by ROTEM results).
  That is, in each case, the same protamine dosage applies to both groups.
Maximal Clot firmness (MCF) | 10 minutes after induction of anesthesia
  CT, CFT, A10, MCF - Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
Maximal Clot firmness (MCF) | 1 minutes after rewarming (during CPB)
  CT, CFT, A10, MCF - Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
Maximal Clot firmness (MCF) | 15 minutes after injection of protamine (after cessation of CPB for reversal of heparin)
  CT, CFT, A10, MCF - Additional parameters assessed by ROTEM (INTEM, EXTEM, FibTEM)
  Dosage of heparin and protamine is only affected by patients' real body weight (not by ROTEM results).
  That is, in each case, the same protamine dosage applies to both groups.
the number of patients who received plasma product transfusion including fresh frozen plasma, cryoprecipitate and platelet concentrate. | postoperative 48 hours for plasma product transfusion
  plasma product transfusion - the number of patients who received plasma product transfusion including fresh frozen plasma, cryoprecipitate and platelet concentrate.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiac Anesthesiology, Department of Anesthesiology and Pain Medicine, Cardiovascular Hospital, Severance Hospital, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided